CLINICAL TRIAL: NCT01456234
Title: Comparison of Time From Symptom Onset to Oseltamivir Access When Oseltamivir is Prescribed by Pharmacists vs. Physicians and the Impact on Symptoms, Oseltamivir Resistance, and Patient Safety
Brief Title: Time to Oseltamivir Access When Prescribed by Pharmacists Versus Physicians (ACCESS)
Acronym: Access
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Trial Management Group Inc. (Network)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CAI-002-11
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with Oseltamivir Prescription (Active Comparator): Patients arriving at the pharmacy with a prescription for Oseltamivir
  Interventions: Drug: Oseltamivir
- Patients with signs, symptoms of flu (Experimental): Patients arriving at the pharmacy with signs, symptoms of flu that the pharmacist diagnoses as having flu and being suitable for pharmacist prescribing of Oseltamivir according to an algorithm.
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Oseltamivir — Oseltamivir 75 mg BID
  Other Names: Tamiflu

SUMMARY:
The main purpose of this study is to see if patients with the flu would receive oseltamivir treatment more quickly if it were prescribed by a pharmacist as compared to a physician, and to see if there is any difference in the effect of treatment on flu symptoms and overall health. Another reason for doing the study is to see how accurately pharmacists can diagnose the flu as compared to physicians. Viruses that are exposed to antiviral medications (like oseltamivir) sometimes develop a resistance to the medication. This means that the medication is no longer as effective in treating the symptoms caused by the virus. The development of viral resistance to oseltamivir will also be followed in this study.

ELIGIBILITY:
Inclusion Criteria Group 1

1. Male and female subjects ≥ 18 years of age presenting at the pharmacy with a current prescription for oseltamivir (75 mg capsule BID for 5 days as per the Canadian label) for the treatment of their own current influenza symptoms
2. Willingness to undergo 2 nasal swab procedures
3. Willingness to participate in the study as evidenced by a written and signed Informed Consent Form

Inclusion Criteria Group 2

1. Male and female subjects ≥ 18 years of age presenting at the pharmacy with indicative clinical symptoms/signs of uncomplicated acute illness due to influenza infection that started within a maximum of 2 days prior to the visit to the pharmacy (see Appendix A:

   FACTSS Influenza Diagnostic Tool)
2. Suitable for oseltamivir treatment at a dose of 75 mg BID (see Appendix B: Algorithm for Determining Suitability of Pharmacist Prescribing of Oseltamivir)
3. Willingness to undergo 2 nasal swab procedures
4. Willingness to pay for (if not covered by insurance) and receive treatment with oseltamivir
5. Willingness to participate in the study as evidenced by a written and signed Informed Consent Form

Exclusion Criteria Group 1

1. Subjects who have been prescribed any other formulation (i.e., oral suspension) or dose regimen of oseltamivir, or any other antiviral medication for the treatment of influenza
2. Individuals presenting at the pharmacy with an oseltamivir prescription who themselves do not currently have a diagnosis of influenza (e.g., individuals filling a prescription for someone else who is currently infected with influenza; individuals filling a prescription that they or someone else will use for prevention of influenza infection or for treatment of a future influenza infection)
3. Subjects who have received an oseltamivir prescription from a physician participating in the study
4. Subjects for whom the oseltamivir prescription is not filled for any reason
5. Subjects who, in the opinion of research personnel, will not comply with the study procedures
6. Staff in the pharmacy or the primary care clinic who are involved in the study, and their family members

Exclusion Criteria Group 2

1. Subjects who have already started treatment with an antiviral medication for their current influenza symptoms
2. Subjects for whom the oseltamivir prescription is not filled for any reason
3. Subjects who, in the opinion of the investigator, are not suitable for the study for clinical or other reasons (e.g., the patient requires hospitalisation or will not be able to comply with study procedures)
4. Staff in the pharmacy or the primary care clinic who are involved in the study, and their family members

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Time from symptom onset to Oseltamivir access | Confirmed at Visit 1, Day 1

SECONDARY OUTCOMES:
Positive Predictive Value (PPV) of Influenza Clinical Diagnosis | Confirmed at Visit 1, Day 1
Oseltamivir Resistance | Confirmed at Visit 1, Day 1 and Visit 2, Day 5
Influenza Signs and Symptoms | Collected from Day 1 to Day 5
Adverse Events | Collected over 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Anil K Gupta, MD, Principal Investigator — Private Practice
Locations (15):
- Canada (15):
  - Paradise Medical Clinic, St. John's, Newfoundland and Labrador
  - Aviva Medical Clinical Trials Group, Burlington, Ontario
  - Co-Medica Research Network, Courtice, Ontario
  - Dr. Sameh Fikry Medicine Professional Corporation, Kitchener, Ontario
  - Schacter Medicine Professional Corporation, London, Ontario
  - Springbank Medical Centre, London, Ontario
  - Taunton Health Centre, Oshawa, Ontario
  - Steeple Hill Medical Centre, Pickering, Ontario
  - London Road Diagnostic Clinic and Medical Centre, Sarnia, Ontario
  - DCTM Clinical Trials Group Ltd., Strathroy, Ontario
  - Dr. Anil Gupta, Toronto, Ontario
  - Source Unique Research, Dollard-des-Ormeaux, Quebec
  - Omnispec Clinical Research Inc., Mirabel, Quebec
  - Metropolitan Clinical Research Centre, Montreal, Quebec
  - ALPHA Recherche Clinique, Québec, Quebec